CLINICAL TRIAL: NCT00830817
Title: A Randomized, Double-Blind Phase I Study to Evaluate Topically Applied WBI-1001 Cream in Patients With Psoriasis.
Brief Title: Double-Blind Study of Topical WBI-1001 Cream on Patients With Psoriasis
Acronym: WBI-1001-101
Status: Completed | Type: Observational
Sponsor: Welichem Biotech Inc. (Industry)
Responsible Party: Robert Bissonnette; Principal Investigator, Innovaderm Research, Inc.,
Other Study IDs: WBI-1001-101; control # 114963
Record Dates: First submitted 2009-01-26; First posted 2009-01-28 (Estimated); Last update posted 2009-01-28 (Estimated); Status verified 2009-01

CONDITIONS: Psoriasis
Keywords: Topical cream application; Mild to moderate psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood plasma samples retained following PK analyses.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to evaluate primarily the safety and tolerability and secondarily the efficacy of topically applied WBI-1001 cream in patients with mild to moderate psoriasis. Double-blind, randomized, placebo controlled study of 36 patients, treated for 28 days plus a 7 day follow-up.in which the patients were divided into six cohorts: Cohort 1 at 0.5% QD;Cohort 2 at 0.5% BID; Cohort 3 at 1.0% QD; Cohort 4 at 1.0% BID; Cohort 5 at 2.0% QD; Cohort 6 at 2.0% BID.Efficacy assessed by PGA,target lesion assessment and BSA. Safety assessed through vital signs, ECG, AEs and Plasma PK via Cmin, Cmax,Tmax and AUCo-t.

DETAILED DESCRIPTION:
Patients initiated screening within 4 weeks of commencing study treatment. Based on progression of the study, at day 0 patients were assigned to one of six treatment Cohorts. Patients were randomized to treat all areas except the face, scalp, groin and genital areas. Patients in Cohort 1 were treated on one side with a thin layer of active cream and the other with placebo; in the absence of significant AEs by 14 days after the last treatment in the Cohort escalation to the next Cohort was allowed, and each Cohort respectively.

During the treatment period patients visited the study centre weekly for safety, tolerability and efficacy assessment. On these study visit days blood draws were done between 7.00 and 10.00am prior to that morning's application of cream.

The study enrolled healthy male and female patients aged 18-65 y.o. with clinical diagnosis of stable plaque psoriasis for >months affecting a maximum of 6% of BSA with a minimum of 0.5% BSA on each side of the body and a minimum of one plaque at least 2x2 cm on each side excluding elbow and knee.

ELIGIBILITY:
Inclusion Criteria:

* PGA score at day 0 must be 2,3 or 4.
* In good overall health.
* Women of child bearing potential to have negative serum beta-human chorionic gonadotropin pregnancy test before randomization
* Must be prepared to use adequate means of contraception
* Must not be lactating.
* Male partners of females in the study must be prepared to use adequate means of contraception.
* Must comply with study protocol and attend all visits.
* Provide written consent prior to participating in the study.

Exclusion Criteria:

* Spontaneously improving or rapidly deteriorating psoriasis.
* Patients with other diseases (especially dermatological, immunodeficiency or neurological/psychiatric) that might interfere with assessment of plaque psoriasis.
* Systemic immunomodulatory therapy in past 36 weeks, phototherapy in past 4 weeks, various psoriatic chemotherapies and beta blockers in the past 2 weeks

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Males and female18-65 yo. inclusive Mild to moderate plaque psoriasis
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2007-07; Primary Completion 2008-04 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Evaluate safety and tolerability of topically applied WBI-1001 cream, and to assess the pharmacokinetics based on plasma concentrations | 35 days

SECONDARY OUTCOMES:
Obtain initial evaluation of efficacy of topically applied WBI-1001 cream in patients with mild to moderate psoriasis. | 35 days

CONTACTS AND LOCATIONS:
Overall Officials: John m Webster, PhD, D.Sc., Study Chair — Welichem Biotech Inc.; Liren Tang, Ph.D, Study Director — Welichem Biotech Inc.
Locations (1):
- Innovaderm Research inc., Montreal, Quebec, Canada